CLINICAL TRIAL: NCT05323110
Title: A Double-blind, Randomized, Placebo-controlled, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of Single- and Multiple-ascending Doses of Intravenously Administered Anti-LIGHT Monoclonal Antibody CBS001 in Healthy Volunteers
Brief Title: Study of Intravenously Administered Anti-LIGHT Monoclonal Antibody CBS001 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Portfolio reprioritization
Sponsor: Capella Bioscience Ltd (Industry)
Collaborators: Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBS001-01
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Chronic Inflammatory Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part A - Cohort 1A (Experimental): Single dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part A - Cohort 2A (Experimental): Single dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part A - Cohort 3A (Experimental): Single dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part A - Cohort 4A (Experimental): Single dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part A - Cohort 5A (Experimental): Single dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part A - Cohort 6A (Experimental): Single dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part A - Cohort 7A (Experimental): Single dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part A - Cohort 8A (Experimental): Single dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part B - Cohort 1B (Experimental): Multiple dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part B - Cohort 2B (Experimental): Multiple dose cohort
  Interventions: Drug: CBS001; Drug: Placebo
- Part A - Cohort 3B (Experimental): Multiple dose cohort
  Interventions: Drug: CBS001; Drug: Placebo

INTERVENTIONS:
Drug: CBS001 — Intravenously administered, humanised anti-LIGHT IgG monoclonal antibody.
Drug: Placebo — CBS001 matched placebo

SUMMARY:
A Phase 1, first in human (FIH), single-centre, double-blind, randomized, placebo-controlled, dose escalating trial to assess the safety and tolerability, pharmacokinetics (PK), immunogenicity and pharmacodynamics (PD) of CBS001 in healthy subjects. The study will be conducted in 2 parts:

Part A: Single ascending intravenous (IV) doses of CBS001 Part B: Multiple ascending IV doses of CBS001

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy volunteer.
2. Aged 18-65 years.
3. A body mass index (BMI; Quetelet index) in the range 18.0-30.9. Body Mass Index = weight (kg)/(height[m]^2
4. Ability to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
5. Willingness to give written consent to participate after reading the information and consent form (ICF), and after having the opportunity to discuss the trial with the investigator or their delegate.
6. Agree to follow the contraception requirements of the trial
7. Agree not to donate blood or blood products during the study and for up to 3 months after the administration of the trial medication or until the final follow-up visit (whichever is longer).
8. Registered with a General Practitioner (GP) in the United Kingdom.
9. Willingness to give written consent to have data entered into The Overvolunteering Prevention System (TOPS).

Exclusion Criteria:

1. Woman who is pregnant or lactating, or pre-menopausal woman who is sexually active and not using a reliable method of contraception.
2. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
3. Isolated bilirubin > 1.5 x upper limit of normal (ULN). Isolated bilirubin > 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35% indicative of Gilbert's syndrome.
4. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
5. Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, allergic diseases such as asthma or atopic dermatitis requiring medication, or history of any psychotic mental illness.
6. Presence or history of severe adverse reaction to any drug or a history of sensitivity to any CBS001 excipient.
7. Use of a prescription medicine (except hormone contraceptives or hormone replacement therapy [HRT] in women) during the 28 days before the (first) dose of trial medication, or use of an over-the-counter medicine (except acetaminophen [paracetamol], dietary supplement, or herbal remedy) including St John's Wort during the 7 days before the (first) dose of trial medication.
8. Receipt of an investigational product (including prescription medicines) as part of another clinical trial within the 3 months before [first] admission to this study; in the follow-up period of another clinical trial at the time of screening for this study.
9. Receipt of an approved or investigational biological product within the 12 months before screening.
10. Receipt of a vaccination (except COVID-19 vaccine) within 28 days before (first) dose of trial medication, or planned vaccination during the study.
11. Presence or history of drug or alcohol abuse, or intake of more than 14 units of alcohol weekly, or more than 10 cigarettes or 6.25 g of tobacco daily.
12. Blood pressure and heart rate in supine position at the screening examination outside the ranges: blood pressure 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40-100 beats/min. Repeat measurements are permitted if values are borderline (ie values that are within 5 mm Hg for blood pressure or 5 beats/min for heart rate) or if requested
13. Corrected QT interval (QTcF) value greater than 450 msec (men) or greater than 470 msec (women) measured on 12-lead ECG at the screening examination. Triplicate measurements will be made, and a mean value used to determine eligibility. A repeat (in triplicate) is also allowed on 1 occasion for determination of eligibility. Participants can be included if the repeat value is within range or still borderline, but deemed not clinically significant by the investigator.
14. Possibility that the volunteer will not cooperate with the requirements of the protocol.
15. Evidence of drug abuse on urine testing.
16. Positive test for hepatitis B, hepatitis C (unless has received curative antiviral treatment and has a negative polymerase chain reaction [PCR] for viral load) or HIV. Loss of more than 400 mL blood during the 3 months before the study, eg as a blood donor.
17. Objection by GP to volunteer entering study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] (Part A) | Up to Day 190
  Number of Participants with One or More Drug Related Adverse Events (AEs) or any Serious AEs
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] (Part B) | Up to Day 247
  Number of Participants with One or More Drug Related Adverse Events (AEs) or any Serious AEs

SECONDARY OUTCOMES:
CBS001 plasma evaluation over time (Part A) | Up to Day 190
  CBS001 plasma concentrations will be measured at specified visits
CBS001 plasma evaluation over time (Part B) | Up to Day 247
  CBS001 plasma concentrations will be measured at specified visits
Antibodies against CBS001 in serum (Part A) | Up to Day 190
  Immunogenicity
Antibodies against CBS001 in serum (Part B) | Up to Day 247
  Immunogenicity

OTHER OUTCOMES:
Serum concentrations of pharmacodynamic marker(s) (Part A) (Exploratory) | Up to Day 190
  Serum concentrations of pharmacodynamic marker(s) will be measured at specified visits
Serum concentrations of pharmacodynamic marker(s) (Part B) (Exploratory) | Up to Day 247
  Serum concentrations of pharmacodynamic marker(s) will be measured at specified visits

CONTACTS AND LOCATIONS:
Locations (1):
- HMR, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No